CLINICAL TRIAL: NCT02236338
Title: Radiofrequency Ablation vs Laser Ablation of the Incompetent Greater Saphenous Vein: A Prospective Randomized Trial
Brief Title: Radiofrequency Ablation vs Laser Ablation of the Incompetent Greater Saphenous Vein
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM11792
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Chronic Venous Insufficiency
Keywords: chronic venous insufficiency; varicose vein; greater saphenous vein
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency Ablation (Active Comparator): Device: ClosureFAST radiofrequency catheter (VNUS Medical Technologies Inc, San Jose, CA).
  Patients will have the intervention, ablation of the incompetent greater saphenous vein, using this device.
  Interventions: Procedure: Ablation of the Incompetent Greater Saphenous Vein; Device: ClosureFAST radiofrequency catheter
- Laser Ablation (Active Comparator): Device: EVLT 980nm diode laser system (Angiodynamics, Queensbury, NY).
  Patients will have the intervention, ablation of the incompetent greater saphenous vein, using this device.
  Interventions: Procedure: Ablation of the Incompetent Greater Saphenous Vein; Device: EVLT 980nm diode laser system

INTERVENTIONS:
Procedure: Ablation of the Incompetent Greater Saphenous Vein — For each patient, the Greater Saphenous Vein (GSV) will be accessed just below the knee. After liberal use of anesthesia, the patient will undergo an ablation of the GSV. Half the patients will have this procedure performed using the Laser Ablation device and half will be treated using the Radiofrequency Ablation device. They will be randomly assigned to treatment.
Device: ClosureFAST radiofrequency catheter
  Arms: Radiofrequency Ablation
Device: EVLT 980nm diode laser system
  Arms: Laser Ablation

SUMMARY:
The aim of this study is to perform a randomized, prospective trial comparing the two current methods of treatment for chronic venous insufficiency, in an effort to evaluate complications and outcomes for each method, and ultimately, to see if one is superior to the other.

DETAILED DESCRIPTION:
Chronic venous insufficiency (CVI) is estimated to affect 25 million Americans. This condition leads to varicose veins, aching, fatigue, swelling, ulcerations, and bleeding in the lower extremities. The most common cause is a refluxing or incompetent Greater Saphenous Vein (GSV). This condition results in pooling of deoxygenated blood in the lower extremities rather than successful transport of the blood back to the heart and lungs. The historical treatment has been to surgically remove or 'strip' the GSV so that blood is rerouted through the healthier deep veins. A less invasive treatment option, Endovenous Thermal Ablation, has emerged over the last decade and has virtually replaced stripping. This involves advancing a catheter under ultrasound guidance through the GSV and then advancing a laser fiber or radiofrequency probe through the catheter. These devices then produce the energy to destroy the vein as the catheters are slowly pulled back. While both radiofrequency ablation and laser ablation are accepted treatments, neither technology has been definitively proved to have fewer complications or superior results. This is in part because very few practices have the ability to make a head to head comparison between the two technologies and must choose one or the other secondary to financial constraints. The aim of this study is to perform a randomized prospective trial comparing the two modalities so that more definitive information to evaluate complications and outcome can be obtained and then recommendations on which, if either, technology is superior can be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic chronic venous insufficiency.
* Patients in whom endovenous thermal ablation is clinically indicate.
* Have previously undergone at least 6 weeks of conservative treatment with compression stockings (unless they have venous ulcers, recurrent phlebitis, or bleeding varices).
* Have venous disease that meets CEAP clinical class 2 through 6.
* Have symptoms secondary to Greater Saphenous Vein insufficiency defined as reverse flow in the saphenous vein >0.5 seconds after calf compression or while standing.

Exclusion Criteria:

* Have previously undergone surgery, EVTA, or phlebectomy in that extremity (exclusive of spider vein injections or other cosmetic surface procedures).
* Have a history of DVT.
* Have a history of hypercoaguability disorder.
* Are pregnant or breastfeeding.
* Are nonambulatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2016-08-11 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Sydnor, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiofrequency Ablation: Device: ClosureFAST radiofrequency catheter (VNUS Medical Technologies Inc, San Jose, CA).
  Patients will have the intervention, ablation of the incompetent greater saphenous vein, using this device.
  Ablation of the Incompetent Greater Saphenous Vein: For each patient, the Greater Saphenous Vein (GSV) will be accessed just below the knee. After liberal use of anesthesia, the patient will undergo an ablation of the GSV. Half the patients will have this procedure performed using the Laser Ablation device and half will be treated using the Radiofrequency Ablation device. They will be randomly assigned to treatment.
  ClosureFAST radiofrequency catheter
- Laser Ablation: Device: EVLT 980nm diode laser system (Angiodynamics, Queensbury, NY).
  Patients will have the intervention, ablation of the incompetent greater saphenous vein, using this device.
  Ablation of the Incompetent Greater Saphenous Vein: For each patient, the Greater Saphenous Vein (GSV) will be accessed just below the knee. After liberal use of anesthesia, the patient will undergo an ablation of the GSV. Half the patients will have this procedure performed using the Laser Ablation device and half will be treated using the Radiofrequency Ablation device. They will be randomly assigned to treatment.
  EVLT 980nm diode laser system
Period: Overall Study
Arm/Group | Radiofrequency Ablation | Laser Ablation
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency Ablation | Laser Ablation | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Median (Full Range); unit: years] | 47 [19 to 86] | 48.5 [23 to 86] | 48 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 77 | 157
  Male | 20 | 23 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 78 | 70 | 148
  Race/Ethnicity: African American | 16 | 18 | 34
  Race/Ethnicity: Hispanic | 3 | 7 | 10
  Race/Ethnicity: Asian | 1 | 3 | 4
  Race/Ethnicity: Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Recurrent Clinical Symptoms of an Incompetent Greater Saphenous Vein After Treatment.
Time Frame: Annual follow up, up to 75 months
Population: The mean long-term followup in the EVLA group was 44 (12-64) months, and the mean long-term follow-up in the RFA group was 42 (12-75) months.
Measure: Number; unit: percentage of total participants
Arm/Group | Radiofrequency Ablation | Laser Ablation
Number analyzed (Participants) | 87 | 89
percentage of total participants | 79.3 | 77.5

2. Secondary Outcome: Incidence Rate of Acute Complications
Description: Number of acute complications at one and 6 weeks post intervention
Time Frame: up to 6 weeks post intervention
Measure: Number; unit: number of complications
Arm/Group | Radiofrequency Ablation | Laser Ablation
Number analyzed (Participants) | 100 | 100
number of complications | 0 | 0

3. Other Pre Specified Outcome: Incidence of Post-procedure Pain
Description: Measured with Visual Analog Scale (VAS), with a range of 1-10 with 10 being the most pain.
Time Frame: During post procedure recovery period in clinic, an expected average of 2 hours after surgery.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Radiofrequency Ablation | Laser Ablation
Number analyzed (Participants) | 100 | 100
units on a scale | 1 [1 to 10] | 3 [1 to 10]

4. Other Pre Specified Outcome: Incidence of Objective Post-procedure Bruising
Description: Measured with bruising scale, with a range of 1-10 with 10 being the most bruising.
Time Frame: During post procedure recovery period in clinic, an expected average of 2 hours after surgery.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Radiofrequency Ablation | Laser Ablation
Number analyzed (Participants) | 100 | 100
units on a scale | 2 [1 to 9] | 3 [1 to 8]

ADVERSE EVENTS:
Arm/Group | Radiofrequency Ablation | Laser Ablation
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes